CLINICAL TRIAL: NCT05578365
Title: Effects of an Online Pilates Protocol in Individuals With Chronic Low Back Pain: Randomized Controlled Trial
Brief Title: Online Pilates in Individuals With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Liane de Brito Macedo, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBPOP22-2
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain; Chronic Pain
Keywords: low back pain; Exercise Movement Techniques; Exercise; Chronic Pain; Telerehabilitation
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (Experimental): Pilates method exercise program, performed online, 8 weeks long, twice a week + information on self-management and pain education once a week.
  Interventions: Other: Pilates method
- Control Group (Active Comparator): Information on self-management of low back pain, pain education, and changes in lifestyle habits once a week during 8 weeks.
  Interventions: Other: Pain education

INTERVENTIONS:
Other: Pilates method — Individuals in the Pilates group will perform specific exercises online. There will be 16 sessions, lasting 60 minutes, with 10 minutes of warm-up, 30 to 40 minutes of exercises focusing on the trunk stabilizers muscles, and 10 minutes of cool-down with relaxation, stretching, or meditation. In addition, the individuals will have access to the same information of the control group.
  Arms: Pilates Group
Other: Pain education — Individuals in the control group will receive information on self-management of low back pain, pain education, and changes in lifestyle habits once a week during 8 weeks.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the effects of the Pilates method, performed online, in individuals with chronic low back pain. This is a randomized controlled trial consisting of two arms.

DETAILED DESCRIPTION:
Low back pain is one of the main causes of disability in the world, and physical inactivity is associated with its development. In this sense, Pilates can be used both in the treatment and preventively for this symptomatology. Thus, the aim of this study is to evaluate the effects of the Pilates method, performed online, in individuals with chronic low back pain. This is a randomized controlled trial involving men and women between 18 and 60 years of age with a history of non-specific chronic low back pain and a minimum pain intensity equal to 3 points on the numeric pain scale. Research participants will perform a pre-intervention (EV1) and post-intervention (EV2) assessment, both online. Pain sensation, functional performance, kinesiophobia and perception of global change will be the outcomes evaluated through the following instruments: Numerical Pain Scale, Roland Morris Questionnaire, Tampa Scale for kinesiophobia and Patient Global Impression of Change Scale. Participants included in the study will be randomized into two groups with separate interventions, both lasting eight weeks: online Pilates group and control group. The control group will receive information about self-management of low back pain, pain education, and changes in lifestyle habits; the Pilates group, besides having access to the same information as the control group, will undergo 16 Pilates sessions performed online (2 times/week). The statistical analysis will be done through the independent t test and the Mann-whitney test to investigate the differences between the groups (Pilates online x control), while the paired t test and the Wilcoxon test will be applied to evaluate the effect of the time variable (Pre x Post), considering a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a history of chronic nonspecific low back pain (for more than 12 weeks) and minimum pain intensity of 3 on numerical pain rating scale.

Exclusion Criteria:

* Symptoms related to serious pathologies (such as fever, changes in sensibility, weight loss, constant pain);
* Recent history of spinal fracture, cancer, inflammatory diseases, nerve root involvement, spinal pathologies (such as ankylosing spondylitis, herniated disc with radiculopathy, advanced osteoporosis, spondylolysis, spondylolisthesis);
* Central neurological diseases (such as Parkinson's and stroke), psychiatric (such as depression or schizophrenia);
* Autoimmune diseases;
* Orthopedic surgery in the last year;
* Severe cardiovascular diseases;
* Decompensated metabolic diseases;
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Pain sensation | Change from baseline in pain sensation at eight weeks after the intervention
  Painful sensation measured by numerical pain rating scale (11 points scale)

SECONDARY OUTCOMES:
Functional performance associated to back pain | Change from baseline in functional performance at eight weeks after the intervention
  Functional performance associated with low back pain measured by Roland Morris Disability Questionnaire (24 items - more items is related to worse disability)
Kinesiophobia | Change from baseline in kinesiophobia at eight weeks after the intervention
  Kinesiophobia measured by Tampa Scale of Kinesiophobia (17 to 68 points)
Patient global impression of change | The Patient global impression of change after eight weeks of intervention
  Patient global impression of change measured by a scale with seven points, where 1 is equal to no change or worse and 7 is much better

IPD SHARING:
Plan to Share IPD: No